CLINICAL TRIAL: NCT04309331
Title: Market Research - Acceptability Trial for a New PKU Amino Acid Based Protein Substitute (Dr Schär Medical Nutrition - Mevalia Amino Acids) Mevalia PKU Motion 10 - Tropical or Red Fruits Mevalia PKU Motion 20 - Tropical or Red Fruits
Brief Title: Market Research - Acceptability Trial for a New PKU Amino Acid Based Protein Substitute
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Schär AG / SPA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Motion1
Record Dates: First submitted 2020-02-13; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: PKU; Phenylketonurias; Inborn Errors of Metabolism; Metabolic Disease
MeSH Terms: conditions — Phenylketonurias; Metabolism, Inborn Errors; Metabolic Diseases | interventions — Motion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PKU Motion (Experimental): amino acid based protein substitute
  Interventions: Dietary Supplement: Motion

INTERVENTIONS:
Dietary Supplement: Motion — Amino acid based protein substitute

SUMMARY:
The aim of this study is to demonstrate that a new protein substitute is acceptable and well tolerated in children with PKU.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU or PKU variant requiring a phenylalanine-free protein substitute
* Subjects who are already taking a phenylalanine-free protein substitute and are willing to try the study product for 7 days
* Patients aged 3 years of age to adulthood
* Written informed consent obtained from parental caregiver

Exclusion Criteria:

* Presence of serious concurrent illness
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.
* Any patients having taken antibiotics over the previous 2 weeks leading up to the study.
* Patients less than 3 years of age.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | 7 days
  Questionnaire detailing any GI symptoms, severity and change from usual
  • The collection of daily data about the gastro-intestinal tolerance of the protein substitute.
Product compliance | 7 days
  Daily questionnaire on amounts offered and amounts actually consumed, compared to recommended amount.
Product palatability | 7 days
  Questionnaire data captured to evaluate taste
Product acceptability | 7 days
  Brief tick-box questionnaire on overall liking and acceptability of product

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham Children's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No